CLINICAL TRIAL: NCT04263194
Title: Novel Tailored Network-based rTMS Treatments in Alzheimer's Disease: an Integrated Multiimaging Approach
Brief Title: Network-based rTMS in Alzheimer's Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: IRCCS Centro San Giovanni di Dio Fatebenefratelli (Other)
Collaborators: I.R.C.C.S. Fondazione Santa Lucia (Other); Ministero della Salute, Italy (Other)
Responsible Party: Principal Investigator, Debora Brignani, Principal Investigator, IRCCS Centro San Giovanni di Dio Fatebenefratelli
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: GR-2016-02364718
Record Dates: First submitted 2020-01-30; First posted 2020-02-10 (Actual); Last update posted 2023-03-13 (Actual); Status verified 2023-03

CONDITIONS: Alzheimer Disease, Late Onset; Alzheimer Disease; Cognitive Deterioration
Keywords: TMS; rTMS; Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Intervention Model Description: After recruitment, patients will be randomized and assigned to one of three rTMS treatments: DMN (N=20), CEN (N=20) or placebo (N=20). The rTMS treatment will consist of 2 phases: an intensive phase and a maintenance phase. The intensive phase will involve 3 weeks of treatment, 5 days per week (15 sessions in total). The maintenance will consist of 1 session of treatment every 2 weeks for 5 months (10 sessions in total). Overall, the patients will undergo 25 sessions of rTMS delivered over 6 months. At baseline (T0), at the end of the intensive phase (T1) and at the end of the maintenance phase (T2) all patients will undergo a clinical and cognitive assessment and a multi-modal imaging data collection.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: The study will be a double blind trial, i.e. both patients and clinicians involved in the assessment will be blind to treatment allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Default Mode Network (DMN) (Experimental): The treatment will consist in the individually tailored stimulation of a DMN node (i.e. left inferior parietal lobe).
  Interventions: Device: rTMS
- Central Executive Network (CEN) (Experimental): The treatment will consist in the individually tailored stimulation of a CEN node (i.e. left dorsolateral prefrontal cortex).
  Interventions: Device: rTMS
- Placebo (Placebo Comparator): The treatment will consist in targeting the upper part of the scalp (i.e. CZ) while using a sham rTMS coil.
  Interventions: Device: Sham rTMS

INTERVENTIONS:
Device: rTMS — 25 min of high frequency (20 Hz) repetitive TMS applied at 100% of resting motor threshold (rMT).
  Arms: Central Executive Network (CEN); Default Mode Network (DMN)
Device: Sham rTMS — Placebo intervention will consist in the same procedure but using a sham rTMS coil.
  Arms: Placebo

SUMMARY:
Severe alterations of brain networks connectivity have been described in Alzheimer's disease (AD). Repetitive Transcranial Magnetic Stimulation (rTMS) has gained evidence as an effective tool to modulate brain networks connectivity, leading to a recovery or reorganization of both local and remote brain regions functionally connected to the stimulated area. The investogators propose an innovative tailored network-based rTMS treatment to ameliorate cognitive symptoms in mild AD, through the boosting of connectivity within brain networks affected by AD pathophysiology. The combination of the proposed intervention with an integrated multi-modal imaging approach will allow to evaluate the neural mechanisms underlying the clinical response to the treatment and to define quantitative markers of clinical impact on AD. If successful, the present proposal would immediately impact on patient's quality of life, with important implications for the time and costs of delivery of rehabilitative services.

DETAILED DESCRIPTION:
Currently, no effective cure is available for Alzheimer's disease (AD). Repetitive Transcranial Magnetic Stimulation (rTMS) has gained increasing attention as a potential treatment for various neurological and psychiatric disorders, but available rTMS studies are flawed by inaccurate anatomical targeting, inadequate sample size, unsatisfactory controls and lacking blindness. To date, the elective target area of rTMS interventions in AD has been the dorsolateral prefrontal cortex (DLPFC), a core area of the Central Executive network (CEN), which plays a key role in regulating executive functions, attention and working memory. While the CEN has recently been described as dysfunctional in AD, AD pathophysiology has been mainly associated with the breakdown of the Default Mode network (DMN) and with structural disconnection of its parietal nodes. The DMN plays a crucial role in episodic memory retrieval and incorporates various brain regions, among which parietal areas are highly connected with the rest of the brain. The present multicenter, double-blind, randomized and placebo-controlled study has the ambition to provide evidence of the efficacy of two tailored network-based rTMS treatments in mild AD, through the enhancement of connectivity of CEN and DMN. Innovative integrated multi-modal imaging investigations will further enrich this proposal allowing to identify quantifiable markers underlying the clinical impact of rTMS on AD.

ELIGIBILITY:
Inclusion Criteria:

* Mini-Mental State Examination score >=16, <=24
* Anti-cholinesterase treatment for at least 3 months prior the start date

Exclusion Criteria:

* Enrollment in other clinical and pharmacological trials
* Previous evidence of any other CNS disorder (e.g. epilepsy, infectious diseases, frontotemporal, Parkinson or Pick's disease)
* History of major psychiatric disorders
* History of alchol or substance abuse
* Stress-related skin problems
* Current consumption of psychiatric medication
* Presence of metal implants or any implanted electronics

Ages: 55 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-03-21 (Actual); Primary Completion 2023-09-21 (Estimated); Study Completion 2024-03-21 (Estimated)

PRIMARY OUTCOMES:
Change in ADAS-Cog scale scores | At baseline (T0), up to 4 weeks (T1), through study completion, an average of 6 months (T2)
  A brief neuropsychological assessment used to assess the severity of cognitive symptoms of dementia

SECONDARY OUTCOMES:
Change in CANTAB battery scores | At baseline (T0), up to 4 weeks (T1), through study completion, an average of 6 months (T2)
  The scores on two tests of CANTAB battery (www.cambridgecognition.com):
  * Change in Associative Learning test (PAL)
  * Change in Spatial Working Memory test (SWM)
Change in brain connectivity | At baseline (T0), up to 4 weeks (T1), through study completion, an average of 6 months (T2)
  TMS-evoked cortical responses (TEPs) will serve as markers of reactivity of the stimulated area as well as markers of the connectivity between targeted cortex and functionally connected areas underlying DMN or CEN.
Change in brain plasticity | At baseline (T0), up to 4 weeks (T1), through study completion, an average of 6 months (T2)
  A theta burst stimulation (TBS) protocol will be used to probe plasticity changes
Change in MRI measures of functional and structural connectivity | At baseline (T0), up to 4 weeks (T1), through study completion, an average of 6 months (T2)

CONTACTS AND LOCATIONS:
Overall Officials: Debora Brignani, Principal Investigator — IRCCS Centro San Giovanni di Dio Fatebenefratelli
Locations (1):
- IRCCS Centro San Giovanni di Dio Fatebenefratelli, Brescia, Lombardy, Italy